CLINICAL TRIAL: NCT02162745
Title: Randomized Controlled Trial to Evaluate the Efficacy of Nasal Irrigation in Infants With Bronchiolitis
Brief Title: Nasal Irrigation in Infants With Bronchiolitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 35/12
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Normal saline solution; Hypertonic solution; Nasal irrigation
MeSH Terms: conditions — Bronchiolitis | interventions — Isotonic Solutions; Sodium Chloride; Hypertonic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Isotonic solution (NaCl 0.9%) (Experimental): Single nasal irrigation with 1 ml of isotonic solution (NaCl 0.9%) per each nostril
  Interventions: Drug: Isotonic solution (NaCl 0.9%)
- Hypertonic solution (NaCl 3%) (Experimental): Single nasal irrigation with 1 ml of hypertonic solution (NaCl 3%) per each nostril
  Interventions: Drug: Hypertonic solution (NaCl 3%)
- Supportive care (No Intervention): Wiping the nose, positioning the child, changing a wet diaper, feeding.

INTERVENTIONS:
Drug: Isotonic solution (NaCl 0.9%)
  Arms: Isotonic solution (NaCl 0.9%)
Drug: Hypertonic solution (NaCl 3%)
  Arms: Hypertonic solution (NaCl 3%)

SUMMARY:
Bronchiolitis is a leading cause of acute illness and hospitalization in the first year of life. Most children with bronchiolitis have mild disease and are managed at home with support from primary care providers, while children with more severe symptoms require supportive therapy with oxygen and fluid administration.

Neonates may be obligate nasal breathers until they are at least 2 months old and nasal obstruction may play a relevant role in respiratory resistances throughout the first months of life, whereas nasal passages may exhibit as much as 50% of the total airway resistance. Some guidelines recommend to clear the nostrils of secretions to improve airway patency but no controlled trial on the efficacy of nasal irrigation in infants with bronchiolitis was carried out.

The aim of this randomized controlled trial is to compare normal saline and hypertonic solution for nasal irrigation versus simple supportive care in infants admitted to Emergency Department with bronchiolitis and mild desaturation.

ELIGIBILITY:
Inclusion Criteria:

* infants <1 year
* diagnosis of bronchiolitis with respiratory distress, rhinitis, cough
* oxygen saturation between 88 and 94%

Exclusion Criteria:

* previous treatments (nasal irrigation or suctioning, oxygen, nebulized drugs, nebulized hypertonic solution, antipyretics up to 6 hours before the study entry, oral steroids at any time before study entry)
* chronic illness

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation (%) | up to 50 minutes after allocation
  Measurement of arterial oxygen saturation (SpO2) of hemoglobin with digital pulse oximeter

SECONDARY OUTCOMES:
Respiratory effort (WARME score) | 5, 15, 20, 50 minutes after allocation
  Evaluation of the respiratory effort using the validated WARME score (evaluation of: 1) respiratory rate; 2) prolonged expiration; 2) wheezing; 3) air exchange; 4) muscle use).

CONTACTS AND LOCATIONS:
Overall Officials: Dino Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Silvana Schreiber, RN, Study Director — IRCCS Burlo Garofolo, Trieste, Italy
Locations (2):
- Italy (2):
  - Pediatria, Azienda Ospedaliera Santa Maria Degli Angeli, Pordenone, Friuli Venezia Giulia
  - Emergency Department, IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia